CLINICAL TRIAL: NCT04322175
Title: Pharmacokinetics and Tolerance of Meloxicam Eye Drops in Healthy Volunteers, a Phase I , Single-dose and Multiple-dose, Open-labeled Clinical Trial
Brief Title: Pharmacokinetic and Tolerance Study of Meloxicam Eye Drops in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLXKDYY
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Tolerance
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose pharmacokinetic test (Experimental): The 72 healthy subjects enrolled were admitted to the trial ward the day before the trial. On the day of dosing, the subjects were given 0.1% meloxicam eye drops once, 1 drop / time.
  Interventions: Drug: Meloxicam
- Multiple dose tolerance test (Experimental): Eight healthy subjects were enrolled in the trial ward the day before the trial. 0.1% meloxicam eye drops were administered 4 times, 1 drop / time, and were administered at 8:00, 12:00, 16:00 and 20:00 daily for 3 consecutive days.
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam — Meloxicam Eye Drops
  Other Names: Mobic

SUMMARY:
The pharmacokinetics, safety, and tolerability of meloxicam eye drops in Chinese healthy volunteers were evaluated to provide a basis for the formulation of a phase II clinical trial dosing regimen for this product. Including pre-tests and formal trials, formal trials include single-dose pharmacokinetics tests and multiple-dose tolerance tests (4 times a day for 3 consecutive days).

DETAILED DESCRIPTION:
Meloxicam eye drops is a new class 2 drug of the country. The main ingredients are meloxicam. The other ingredients are hydroxypropyl-β-cyclodextrin, sodium hydroxide, boric acid, sodium chloride and water for injection. Among them, hydroxypropyl-β-cyclodextrin can increase the solubility of meloxicam and improve the stability of the solution. The indication of meloxicam eye drops is non-infectious ocular inflammation, especially for inflammation and complications after cataract surgery. The possible adverse reaction is transient tingling in the eye after eye drops.

Meloxicam is a non-steroidal anti-inflammatory drug (NSAIDS) that selectively inhibits COX-2 cyclooxygenase. It is currently widely used in the treatment of acute and chronic inflammation and pain, and its mechanism of action is to prevent the production of prostaglandins (PGs) that cause inflammation by inhibiting cyclooxygenase (COX). Non-infectious ocular inflammation is usually caused by the synthesis and release of inflammatory mediators such as prostaglandin (PG) after eye tissues are stimulated. Because non-steroidal anti-inflammatory drugs have anti-inflammatory, anti-allergic and analgesic effects, and have no adverse effects of glucocorticoids, their application in ophthalmology has been valued.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this trial and sign the informed consent before the trial;
* Age: 18 to 45 years old (including 18 and 45 years old) healthy subjects, both male and female;
* Weight and body mass index: female subjects weigh ≥45.0kg and male subjects weigh ≥50.0kg,BMI is in the range of 19 ～ 26 kg / m2 (including 19 and 26);
* Physical examination, vital signs, laboratory examination and ECG examination during the screening period are normal or different Often without clinical significance;
* The corrected visual acuity of both eyes should be ≥1.0. The intraocular pressure, slit lamp, and fundus examination are normal or abnormal. It has no clinical significance. The target eye SchirmerⅠ test result during the screening period is ≥10 mm;
* Subjects were able to communicate well with the researcher and understood and were willing to comply with the requirements of this study.

Exclusion Criteria:

* Allergic constitution, allergic diseases or known allergies to research drugs / similar drugs;
* Past or current suffering from circulatory system, respiratory system, digestive system, blood system,Menstrual system, immune system, urinary system, endocrine system, and mental illness may be significant Any condition that affects the absorption, distribution, metabolism, and excretion of the drug or affects the safety of the subject;
* People with eye diseases, including history of internal eye surgery or laser surgery;
* Infection screening is abnormal and clinically significant;
* Used any medicine in the last 2 weeks;
* Underwent surgery within 4 weeks prior to the trial, or plan to perform surgery within 2 weeks of the end of the study surgeon;
* Those who need to wear contact lenses during the trial;
* A history of substance abuse, or a positive urine test for substance abuse(Ketamine, morphine, methamphetamine, dimethylene oxyamphetamine, tetrahydrocannabinol);
* Women with a positive blood pregnancy test; women who have not taken effective contraception in the last month,Pregnant and lactating women; women and men of childbearing age who cannot take effective contraception during the trial and within six months after the trial is over;
* Smokers and alcoholics (smokers on average more than 5 cigarettes / day, alcohol consumption on average 2 units / day, 1unit = 10 mL of ethanol, ie 1 unit = 200 mL of beer with 5% alcohol or 25mL of white wine with 40% alcohol or 83mL of wine with 12% alcohol) or a positive breath test, or during the study Stop using any tobacco products and not stop alcohol intake;
* Those who donated more than 200 mL of blood in the 90 days before the test, or lost blood of more than 200 mL for other reasons;
* Participants in any other clinical trials within 90 days before screening;
* Subjects refused to discontinue any use of methyl groups 48 hours before the end of the study until the end of the study xanthine drinks or foods, such as caffeine (coffee, tea, cola, chocolate, etc.), and beverages containing grapefruit;
* Any other condition that the investigator considers inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of drug prototype-meloxicam in tears of each subject, ng · h / ml | 2 days
  In a single administration test, tear samples were collected 0.5, 1, 2, 4, 6, 8, 10, 12 and 24 hours after administration, and 8 eyes were taken at each time point.LC-MS
Intraocular pressure examination,mmHg | 1 day
  In the multiple dose tolerance test, IOP was performed 2 hours (± 20min) after the second dose of Day2.
Corneal fluorescence staining,levels | 3 days
  Corneal fluorescence staining during the multiple dose tolerance test (Day1-Day3) 1 h after the last daily dose (time window ± 10 min).

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Ph.D., Principal Investigator — Beijing Tongren Hospital, Capital Medical Univsersity
Locations (1):
- Institution of Drug Clinical Trials, Beijing, Beijing Municipality, China